CLINICAL TRIAL: NCT03746158
Title: University of Massachusetts Amherst
Brief Title: Interindividual Variation in Excretion of Curcumin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-4937
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-03

CONDITIONS: Metabolites; Gut Microbiota
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Curcumin (Experimental): subjects will be assigned to consume one capsule of curcumin (330 mg of curcumin per capsule) three times a day (one capsule with each meal).
  Interventions: Dietary Supplement: curcumin

INTERVENTIONS:
Dietary Supplement: curcumin — subjects will be assigned to consume one capsule of curcumin (330 mg of curcumin per capsule) three times a day (one capsule with each meal).

SUMMARY:
The objective of this project is to elucidate the interindividual variations in excretion of curcumin and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 year old healthy adults

Exclusion Criteria:

* Exclusion criteria included those who are <18 or >30 years old, have a BMI of <20 or >29 kg/m2, have a weight change >4.5 kg in the past 3 months, exceed exercise activities of a curcumin level over the past 3 months, have any diseases, especially intestinal disorders, had abnormal liver or kidney function tests. Those who smoke, consume more than two alcoholic drinks per day, use medication affecting gut microbiota profile (e.g., antibiotics and probiotics) in past three months will also be excluded.
* Additionally, this study excludes menopausal women, those using hormone-based contraceptives, those with abnormal menstrual cycles, and those who are pregnant, lactating or planning to become pregnant.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Determine the concentration of curcumin and its metabolites in the human fecal samples. | 3-4 weeks
  Utilize LC-MSMS to identify and quantify the curcumin and its metabolites in the subjects fecal samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Applied Life Sciences, Amherst, Massachusetts, United States